CLINICAL TRIAL: NCT06600087
Title: Long-term Evolution of Risky Sexual Behaviors and Prevalence of Sexually Transmitted Infections Among Pre-Exposure Prophylaxis Users: A Retrospective Observational Study in Gironde, France
Brief Title: Exploring Long-term Risks and STI Prevalence in Pre-Exposure Prophylaxis Users in Gironde, France
Acronym: SAFER-PrEP
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2024/03
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: HIV Infections; Sexually Transmitted Diseases
Keywords: Pre-Exposure Prophylaxis; HIV Prevention; Sexually Transmitted Infections; Long-term Effects; Behavioral Trends
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PrEP less than a year
  Interventions: Behavioral: Questionnaire
- PrEP for over a year
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Standardized self-administered questionnaire specifically designed for this study.

SUMMARY:
SAFER-PrEP investigates the long-term impact of Pre-Exposure Prophylaxis (PrEP) on risky sexual behaviors and Sexually Transmitted Infection (STI) prevalence among users in Aquitaine. The study aims to compare STI rates over the last three months between individuals on PrEP for over a year and those on PrEP for less than a year. This retrospective observational research offers insights into the evolving dynamics of sexual health practices, informing future PrEP prescriptions and enhancing preventive strategies.

DETAILED DESCRIPTION:
Scientific Rationale: The SAFER-PrEP study stems from the imperative to comprehend the intricate interplay between Pre-Exposure Prophylaxis (PrEP) utilization and sexual health dynamics. Amidst the increasing adoption of PrEP for HIV prevention, concerns arise regarding potential behavioral shifts and heightened risks for Sexually Transmitted Infections (STIs). The comprehensive investigation into these phenomena seeks to provide nuanced insights into the long-term implications of PrEP, contributing valuable data to public health initiatives and refining prevention strategies in the face of evolving sexual health landscapes.

Procedure: Participants, comprising individuals on PrEP for over a year and those for less than a year, will be engaged through a observational approach. Data will be collected via self-administered questionnaires during routine consultations for PrEP renewal in various medical settings, including hospitals and private practices. This comprehensive strategy enables a nuanced exploration of sexual behaviors and STI prevalence.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years old;
* Participants using PrEP for at least 6 months ;
* French-speaking, without comprehension disorders ;
* being affiliated to health insurance ;
* Willing to participate and to sign informed consent.

Exclusion Criteria:

* Individuals with known HIV positivity;

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants on Pre-Exposure Prophylaxis (PrEP) for HIV
Sampling Method: Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2025-06-03 (Actual)

PRIMARY OUTCOMES:
Prevalence of Sexually Transmitted Infections (STIs) within the last three months | At baseline (Day 0)

SECONDARY OUTCOMES:
Prevalence of risky sexual behaviors in the last three months. | At baseline (Day 0)
Description of the population of PrEP users in Aquitaine. | At baseline (Day 0)
Behavioral trends in PrEP users based on self-administered questionnaires. | At baseline (Day 0)
Comparison of STI prevalence between PrEP users for over a year and those for less than a year. | At baseline (Day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe JOSEPH, Prof, Principal Investigator — jean-philippe.joseph@u-bordeaux.fr
Locations (8):
- France (8):
  - Cegidd de Bordeaux, Bordeaux
  - CHU de Bordeaux - Service de médecine interne et maladies infectieuses, Bordeaux
  - Maison de la Santé de l'Hôpital Saint-André - Médecine Générale, Bordeaux
  - Cabinet de Medecine Generale, Fargues-Saint-Hilaire
  - Cabinet de Medecine Generale, Le Teich
  - Cegidd de Libourne, Libourne
  - Cabinet de Medecine Generale, Mérignac
  - Cegidd de Perigueux, Périgueux

IPD SHARING:
Plan to Share IPD: No